CLINICAL TRIAL: NCT04914390
Title: A Prospective, Open, Single-arm, Phase Ⅱ Clinical Study of Anlotinib Combined With Tislelizumab and AT in the Neoadjuvant Treatment of Triple-negative Breast Cancer
Brief Title: A Phase Ⅱ Study of Anlotinib Combined With Tislelizumab and AT in the Neoadjuvant Treatment of Triple-negative Breast Cancer
Acronym: NeoATCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Luojing, Prof., Sichuan Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTERBC008
Record Dates: First submitted 2021-05-31; First posted 2021-06-04 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Triple-negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — tislelizumab; anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab + Anlotinib + Chemotherapy (Experimental): Participants receive Tislelizumab every 3 weeks (Q3W) + Anlotinib d1-14 (Q3W) + AT regimen (Q3W) x 6 cycles as neoadjuvant therapy prior to surgery.
  Interventions: Drug: AT regimen; Drug: Tislelizumab; Drug: Anlotinib

INTERVENTIONS:
Drug: AT regimen — Doxorubin 60mg/㎡ d1 or Epirubicin 75mg/㎡ d1 and Nab-paclitaxel 260mg/㎡ d1 of Cycles 1-6 (Q3W) of the neoadjuvant phase of the study; IV injection.
  Other Names: Anthracycline/Nab-paclitaxel
Drug: Tislelizumab — 200mg on d1 of Cycles 1-6 (Q3W) of the neoadjuvant phase of the study; IV injection.
  Other Names: BGB-A317
Drug: Anlotinib — 8mg on d1-14 of Cycles 1-5 (Q3W) of the neoadjuvant phase of the study; po. Arotinib is a small molecule multi-target TKI, which exerts its effect by inhibiting angiogenesis, a critical component of tumour growth and metastasis.
  Other Names: AL3818

SUMMARY:
This is a prospective, single-arm and open-label phase II study, evaluating the efficacy and safety of anlotinib combined with tislelizumab and AT regimen as neoadjuvant treatment for triple-negative breast cancer. Participants will undergo/receive PDL1 testing after enrollment. All patients will be receive 6 cycles of low-dose anlotinib combined with tislelizumab and AT（Doxorubicin or Epirubicin+albumin-bound paclitaxel）regimen, followed by surgery.

ELIGIBILITY:
Inclusion Criteria:

* Has newly diagnosed, locally advanced TNBC, as defined by the most recent American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines.
* Age 18-75 years, female patients
* ECOG performance status ≤1
* Has previously untreated locally advanced non-metastatic (M0) TNBC defined as the following combined primary tumor (T) and regional lymph node (N) staging per current American Joint Committee of Cancer (AJCC) staging criteria for breast cancer as assessed by the investigator based on radiological and/or clinical assessment:T1c, N1-N2、T2, N0-N2、T3, N0-N2、T4a-d, N0-N2
* Demonstrates adequate organ function:

  1. Patients did not receive blood, platelet transfusion or growth factor support treatment within 14 days before blood sample collection in the screening period, and needed to meet:

     1. Hemoglobin（HB）>= 9g / dL;
     2. The absolute value of neutrophil（ANC）>= 1.5 x 10^9/L;
     3. Platelets（PLT）>= 100 x 10^9/L;
  2. The biochemical inspection must meet the following indicators:

     1. Serum creatinine（Cr）<= 1.5 ULN, or creatinine clearance（CCr）>= 60mL / min;
     2. Total bilirubin（TBIL）<= 1.5 ULN, Or total bilirubin>1.0 ULN but direct bilirubin <= 1.0 ULN;
     3. AST and ALT <= 2.5 ULN.
* Female participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through >= 120 days after the last dose of study treatment, and have a negative serum pregnancy test <= 7 days before the first administration of the study drug.

Exclusion Criteria:

* Has a history of invasive malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
* Has received prior chemotherapy, targeted therapy, and radiation therapy within the past 12 months.
* Has received prior therapy with an anti-programmed cell death protein 1 (anti-PD-1), anti-programmed death - ligand 1 (anti-PD-L1), or antiangiogenic drug therapy.
* Patients who are known to be allergic to Tislelizumab, Anlotinib, nab-paclitaxel or Anthracyclines;
* Has multiple factors affecting oral medication. Such as inability to swallow, chronic diarrhea and intestinal obstruction;
* Patients with any severe and/or uncontrolled disease, including:

  1. Patients whose blood pressure control is not ideal (systolic pressure >= 150 mmHg, diastolic pressure >= 100 mmHg);
  2. Having grade I or above myocardial ischemia or infarction, arrhythmia (including QTc >= 450ms(male) or QTc >= 470ms(female) and grade >= 2 congestive heart failure (New York Heart Association (NYHA) classification);
  3. Active or uncontrolled severe infection;
  4. Antiviral treatment for cirrhosis, decompensated liver disease, active hepatitis or chronic hepatitis;
  5. Renal failure requires hemodialysis or peritoneal dialysis;
  6. A history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or a History of organ transplantation;
  7. Poor control of diabetes mellitus (FBG) > 10mmol/L;
  8. Urine routine indicated urinary protein >= ++, and confirmed 24-hour quantitative urinary protein > 1.0g;
  9. Patients with epileptic seizures requiring treatment;
* Patients whose tumors have invaded around important blood vessels according to imaging findings or whose tumors are likely to invade important blood vessels or whose tumors are obviously necrotic and cause fatal massive hemorrhage according to the judgment of the researchers during the follow-up study;
* Patient has experienced A number of thrombosis events, such as cerebrovascular accident (including temporary ischemic attack), deep vein thrombosis and pulmonary embolism within 6 months;
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months;
* Regardless of the severity, patients with any physical signs or history of bleeding, patients with bleeding or bleeding events greater than or equal to CTCAE 3 within four weeks prior to the first administration, or patients with unhealed wounds, fractures, gastric and duodenal active ulcers, ulcerative colitis, or unresected tumors have active bleeding, or may be caused as determined by the researchers. Other conditions of gastrointestinal bleeding and perforation;
* Uncontrolled pleural effusion, pericardial effusion and peritoneal effusion requiring repeated drainage;
* Patients who have participated in clinical trials of other drugs within 4 weeks; Concomitant diseases that, according to the investigator's judgment, may seriously endanger the patient's safety or affect the patient's completion of the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate using the definition of ypT0/Tis ypN0 (i.e., no invasive residual in breast or nodes; noninvasive breast residuals allowed) at the time of definitive surgery | up to approximately 21-24 weeks
  pCR rate (ypT0/Tis ypN0) is defined as the percentage of participants without residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy by current American Joint Committee on Cancer (AJCC) staging criteria assessed by the local pathologist at the time of definitive surgery.

SECONDARY OUTCOMES:
Event-free Survival (EFS) as assessed by Investigator | Up to approximately 3 years
  EFS is defined as the time from randomization to any of the following events: progression of disease that precludes surgery, local or distant recurrence, second primary malignancy (breast or other cancers) or death due to any cause.
pCR rate using an alternative definition, ypT0 ypN0 (i.e., no invasive or noninvasive residual in breast or nodes) at the time of definitive surgery | up to approximately 21-24 weeks
  pCR rate (ypT0 ypN0) is defined as the percentage of participants without residual invasive and in situ cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy by current AJCC staging criteria assessed by the local pathologist at the time of definitive surgery in all participants and in participants with tumors expressing Programmed Death-Ligand 1 (PD-L1).
pCR rate using an alternative definition, ypT0/Tis (i.e., absence of invasive cancer in the breast irrespective of ductal carcinoma in situ or nodal involvement) at the time of definitive surgery | up to approximately 21-24 weeks
  pCR rate (ypT0/Tis) is defined as the percentage of participants without invasive cancer in the breast irrespective of ductal carcinoma in situ or nodal involvement following completion of neoadjuvant systemic therapy by current AJCC staging criteria assessed by the local pathologist at the time of definitive surgery in all participants and in participants with tumors expressing PD-L1.
invasive disease-free survival(IDFS) | up to approximately 3 years
  The time from surgery to the first documented occurrence of an event defined as ipsilateral invasive local recurrence, ipsilateral locoregional invasive recurrence, distant recurrence, contralateral invasive breast cancer, or death from any cause
Overall survival (OS) | up to approximately 5 years
  OS is defined as the time from randomization to death due to any cause. Participants without documented death at the time of the analysis will be censored at the date of the last follow-up.
Percentage of participants who experience an adverse event (AE) | up to approximately 60 weeks
  An AE is defined as any untoward medical occurrence in a participant administered study treatment which does not necessarily have to have a causal relationship with this treatment. An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study treatment or protocol-specified procedure, whether or not considered related to study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of study treatment, is also an AE.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Luo, Prof., Principal Investigator — Sichuan Provincial People's Hospital
Locations (1):
- Department of breast surgery, Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No